CLINICAL TRIAL: NCT04914078
Title: Exacerbations of Severe Asthma in Patients Treated With Mepolizumab: Assessment of Biomarkers and Identification of Biologic Clusters
Brief Title: Severe Asthma Exacerbations and Mepolizumab Treatment
Acronym: ESAM-BIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Alberto Papi, MD, Professor, Università degli Studi di Ferrara
Other Study IDs: 82/2021/Oss/AOUFe - ESAMBIO
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Severe Asthma
Keywords: asthma; exacerbations; eosinophils; infections; mepolizumab
MeSH Terms: conditions — Asthma; Infections | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mepolizumab treated patients: Severe eosinophil severe asthmatic patients treated with anti IL-5 monoclonal antibody Mepolizumab
  Interventions: Drug: Mepolizumab 100 MG

INTERVENTIONS:
Drug: Mepolizumab 100 MG — The patients will treated with subcutaneous Mepolizumab at 100 mg every 30 days. Patients will be recruited among those eligible to Mepolizumab treatment according to the Italian Medicine Agency (AIFA; Agenzia Italiana del Farmaco) guidelines who will accept to participate to the study. In particular inclusion criteria will be: severe (Step 4 and 5 GINA) asthma with at least blood eosinophilic count above 300 cells/mcl at least once in the previous year and ≥150 cells/mcl in the absence of systemic corticosteroid treatment before biological treatment initiation. In addition, one of the following conditions will be required: 1) ≥2 exacerbations in the previous year despite appropriate inhaled treatments or 2) the need for systemic corticosteroids on top of inhaled treatment for at least 6 months in the previous year.

SUMMARY:
This is a hypothesis-generating project to investigate a) infective etiology and b) inflammatory profile of the exacerbations of asthma in severe asthmatic patients treated with the humanized monoclonal antibody against interleukin-5 Mepolizumab. Under these treatment conditions the study will inform on the relationship between these two axes: infection & innate immunity Vs inflammatory profile changes occurring during exacerbation events.

In addition, the study will also explore the effect of Mepolizumab treatment on airway microbial composition and on airway/systemic immune response both at stable state and at the exacerbation.

DETAILED DESCRIPTION:
Longitudinal, observational study to evaluate the infective etiology and the inflammatory profile of asthma exacerbations in severe asthmatic patients treated (as part of routine medical care) with the humanized monoclonal antibody against interleukin-5 Mepolizumab.

The participants receive Mepolizumab as part of routine medical care (see inclusion criteria). The study will assess the effect of the intervention (Mepolizumab) on airway microbial compositions and on airway/systemic inflammation at exacerbation and at stable state.

The patients will be evaluated at baseline (the day of Mepolizumab initiation, before Mepolizumab administration - V0), at 1 month after Mepolizumab initiation (treatment visit - V1), at exacerbation (exacerbation visit - V2) and at 3 months after the exacerbation event (convalescence visit - V3) up to 12-month study period (Table 1). To perform the convalescence visit, a 3-month extension of the study period will be applied if the exacerbation occurs from month 9 to month 12 from the initiation of Mepolizumab. Recurrent exacerbation events will be evaluated separately when a paired-3-month convalescence visit can be performed within the study period.

The patients will contact the center/researchers in case of worsening of the respiratory symptoms to schedule the exacerbation visit. The visit will be performed within 7 days from the beginning of the deterioration of the symptoms.

At each visit, the following procedures will be performed in all the patients: 1) Clinical/pharmacological assessment (including assessment of asthma control; and measurements of central and peripheral fractional exhaled nitric oxide); 2) lung function tests (including lung volumes evaluation and small airway functional assessment by impulse oscillometry - IOS); 3) blood and sputum differential inflammatory cell counts; 4) sputum samples for microbiological assays (conventional sputum cultures and Multiplex Real Time PCR for virus and bacterial detection); 5) blood and sputum samples for cytokine profiling.

In a representative subgroup of patients (n=30) breath condensate, blood and sputum samples will be performed for: 1) airway microbiome (16S ribosomal RNA Sequencing) evaluation; 2) blood innate immune responses; 3) transcriptomics and proteomics of sputum inflammatory cells; 4) breathomics.

The study has been submitted for approval to the ethics committee, and informed written consent will be obtained from each enrolled subject.

ELIGIBILITY:
The cohort of patients included in the study will consist of severe asthmatic patients receiving Mepolizumab as part of routine medical care, i.e. eligible for Mepolizumab treatment according to the Italian Medicine Agency (AIFA; Agenzia Italiana del Farmaco). The patients will receive Mepolizumab treatment irrespective of the enrollment in the study but because of the clinical indication.

Inclusion criteria:

* severe asthmatic patients according to GINA document (Step 4 and 5 GINA)
* blood eosinophilic count above 300 cells/mcl at least once in the previous year and ≥150 cells/mcl in the absence of systemic corticosteroid treatment before biological treatment initiation.
* In addition, one of the following conditions will be required: 1) ≥2 exacerbations in the previous year despite appropriate inhaled treatments or 2) the need for systemic corticosteroids on top of inhaled treatment for at least 6 months in the previous year.

Exclusion criteria:

* COPD
* Active smoking
* Chronic interstitial lung diseases
* Systemic corticosteroid/immunosuppressive treatments for concomitant conditions other than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe eosinophils asthmatic patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Inflammation | 1 year
  Co-primary measurements will be: i) changes in blood and sputum eosinophil counts at exacerbation compared to stable state
Infections | 1 year
  Co-primary measurements will be: ii) changes in the frequency of microbial agent detection in sputum samples at exacerbation compared to stable state.

SECONDARY OUTCOMES:
Lung function FEV1 l | 1 year
  FEV1 litre
Lung function FEV1 % | 1 year
  FEV1% predicted
Lung function FVC l | 1 year
  FVC litre
Lung function FVC % | 1 year
  FVC % predicted
Lung function VC l | 1 year
  vital capacity (VC) litre
Lung function VC % | 1 year
  vital capacity (VC) % predicted
Lung function - Impulsed Oscillometry kPa | 1 year
  R5-R20 (kPa/L/s)
Lung function - Impulsed Oscillometry % | 1 year
  R5-R20 % predicted
Asthma control questionnaire (ACT) | 1 year
  Score ranging from 5 to 25
Fractional exhaled nitric oxide (FeNO) | 1 year
  parts per billions (ppb) in the exhaled breath
Sputum Quantitative bacteriology | 1 year
  Serial dilutions (up to 10-12) of sputum samples will be made and cultured on the appropriate media. Colony- forming units (CFU)/mL will be calculated.
Sputum virus profiling | 1 year
  The commercially available multiplex PCR assay RespiFinder RG® (Qiagen) was used according to manufacture instructions for the simultaneous detection and differentiation of 21 respiratory pathogens, including both viruses and atypical bacteria
Cytokines | 1 year
  cytokines profiling (Th1/Th2/Th17 - pg/ml) in blood serum and sputum supernatants will be assessed by by multiplex immunoassay-based (EMD Millipore Burlington, MA, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No